CLINICAL TRIAL: NCT05933161
Title: GLYcemic Control Evaluation by Continuous Glucose Monitor Compared With a1C in Left Ventricular Assist Device-supported Patients (GLYCEM1C-LVAD)
Brief Title: A Study of Glycemic Control in Left Ventricular Assist
Acronym: GLYCEM1C-LVAD
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Andrew N Rosenbaum, Principal Investigator, Mayo Clinic
Other Study IDs: 22-011965
Record Dates: First submitted 2023-06-28; First posted 2023-07-06 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes Mellitus; Hyperglycemia; Hypoglycemia
Keywords: Left Ventricular Assist Device (LVAD)
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia; Hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Left Ventricular Assist Device (LVAD) supported Type 2 Diabetes Mellitus (T2DM) Subjects: Subjects diagnosed with T2DM who have a LVAD will be provided a Freestyle Libre 3 CGM.
  Interventions: Device: Freestyle Libre 3 Continuous Glucose Monitor (CGM)

INTERVENTIONS:
Device: Freestyle Libre 3 Continuous Glucose Monitor (CGM) — Subjects will be provided a Freestyle Libre 3 CGM for monitoring of blood glucose levels throughout participation in the study (approximately 3 months). CGM data will be uploaded to the LibreLink app on a weekly basis for review of glucose control and consultation with a diabetes-trained provider for any values outside of normal ranges. Adjustments to diet and medication therapy (antihyperglycemic therapy) will be made during consultations to improve episodes of hypoglycemia or severe hyperglycemia that were observed.

SUMMARY:
The study is being conducted to understand if the hemoglobin A1c, a measurement of control of blood sugars over a 3-month time, is valid in patients with Left Ventricular Assist Devices (LVADs) in place. To understand whether it is an adequate measurement, the investigators will compare the A1c to results from a continuous glucose monitor (CGM) measurement of blood sugars. By monitoring blood sugars continuously, the investigators will also assess whether they can get better control of blood sugars with a CGM, including avoiding low blood sugars.

ELIGIBILITY:
Inclusion Criteria:

* Prior implantation of contemporary, centrifugal flow LVAD (HeartWare or HeartMate 3) at any time after 2010
* Diagnosis of type II diabetes mellitus
* Any antihyperglycemic regimen
* Greater than 3 months out from LVAD implantation
* Capable of utilizing smartphone device for LibreLink app for uploading glycemic data
* Patients may be enrolled who have preexisting CGM in place.

Exclusion Criteria:

* Type I diabetics
* Unable to return at 3 month evaluation
* Unwillingness to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with Type 2 Diabetes Mellitus who have a Left Ventricular Assist Device (LVAD) will be recruited from the LVAD clinic at Mayo Clinic in Rochester, MN.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Average glucose values based on continuous glucose monitoring | 3 months
  Average level of blood sugar reported in mg/dL obtained via the Freestyle Libre 3 CGM over a 3 month period.
Estimated average glucose (eAG) values based on hemoglobin-A1c lab values | 3 months
  Estimated average level of blood sugar reported in mg/dL based on conversion of hemoglobin-A1c lab values (eAG=28.7*A1C - 46.7) collected at the 3-month visit.
Estimated average glucose (eAG) values based on fructosamine lab values | 3 months
  Estimated average level of blood sugar reported in mg/dL based on conversion of fructosamine lab values (eAG= 28.7*(0.017 x fructosamine + 1.61) - 46.7) collected at the 3-month visit.

SECONDARY OUTCOMES:
Number of adjustments of antihyperglycemic agents | 3 months
  Number of adjustments made to diet and medication therapy based on consultation from a trained diabetes specialist to improve episodes of hypoglycemia or severe hyperglycemia following review of glucose levels obtained via the Freestyle Libre 3 CGM.
Number of hypoglycemic unawareness episodes | 3 months
  Number of hypoglycemia unawareness episodes defined as periods where subjects did not know that they had low blood sugar according to Freestyle Libre 3 CGM generated alerts.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Rosenbaum, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No